CLINICAL TRIAL: NCT02305004
Title: INTOx A Prospective Measurement of Serum Concentrations of Routine Drugs in Patients Treated in the Intensive Care Unit-A Quality Measurement/Improvement for Clinical Treatment and Forensic Assessment
Brief Title: Blood Serum Concentrations of Routine Drugs in Patients Treated in the Intensive Care Unit.
Acronym: INTOx
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Forensic Toxicology Laboratory, Sweden (Other)
Responsible Party: Sponsor
Other Study IDs: INT001
Record Dates: First submitted 2014-11-27; First posted 2014-12-02 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Serum Concentrations; Intoxication; Post Mortem Concentrations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To follow up the result of a quality measurement based on the results of a new routine for drug analysis introduced during a period of time in the intensive care unit. To ensure the quality of the dose regimen of routine drugs for sedation and analgesics. The aim is also to find out if the routine analysis can give information about if the self- intoxicated patients have taken drugs that were primarily not suspected.To know the serum concentrations of routine drugs in patients who died and will undergo autopsy.

DETAILED DESCRIPTION:
Patients treated in the intensive care unit (ICU) are treated with a variety of sedative and analgesic drugs to be able to undergo intensive care. The amount of drugs that each patient receives is based on standard dosages where the dose regimen is based on clinical studies with a limited number of patients included. Most patients treated in the intensive care unit have a varying degree of cardiac, renal or liver failure which affects the metabolism of the drugs administered. Possibly, the drug concentrations achieved with the standard dosages administered to these patients can vary significantly between patients. This may possibly lead to an extended stay at the ICU which gives the patient an unnecessary suffering, affects the patient's family and increases the cost of health care.

Intoxications due to suicidal purposes is common and usually results in intensive care for those who survive. It is often unknown what type of medication or drugs these patients have been taken and what serum concentration it may result in. Screening methods are available but the information it gives us today may not be enough for the initial acute care of the patient. Also, there are no previous studies with reliable documentation regarding the drug concentrations in the blood of patents that die in the intensive care unit. It is also unknown what kind of drugs and amount of doses given before the death of these patients. It is of significant importance to increase the knowledge in this area to be able to evaluate if the medicines administered before death of patients in intensive care could affect the outcome.

Blood samples will be taken according to routine procedures upon the patients arrival at the ICU and then 2 times per day.

The drug analysis includes drugs used for sedation and analgesia. These samples will be analysed at the national board of forensic medicine (Rättsmedicinalverket) in Linköping. There will also be a screening of unknown or suspected drugs taken by self- intoxicated patients. Sedation ratio by the Richmond agitation sedation scale (RASS) will be evaluated and recorded 3 times per day. An assessment of the visual analogy scale (VAS) will be done for the patients who are awake and are able to cooperate. All physiological measurements will be measured and documented according to local routines. For patients who die at the ICU and undergo autopsy, blood samples will be taken after death for analysis of routine drugs.

ELIGIBILITY:
Inclusion Criteria:

All patients except for children under the age of 7 treated in the Central intensive care unit at Uppsala university hospital, Uppsala Sweden.

Exclusion Criteria:

Age < 7 years old.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients except children under the age of 7 admitted in the ICU at Uppsala University hospital within the time period of 2 years. Estimated number of patients is approximately 1000-1500 patients. The inclusion of patients undergoing autopsy will be after consent from family is obtained according to local routines. Patients undergoing forensic autopsy will also be included in compliance with current regulations. The number of patients in the autopsy group is estimated to be around 100 patients.
Sampling Method: Probability Sample
Enrollment: 359 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Drug serum concentrations inhospital patients at ICU and after death | 1-2 years
  Drug serum concentrations of sedative and analgesics in relation to the quantity of drugs administered and in relation to routine assessment scales of sedation and estimated pain.

SECONDARY OUTCOMES:
Concentrations in relation to organ failure. | 1-2 years
  Drug serum concentration in relation to organ failure.
self intoxicated patients | 1-2 years
  Drug serum concentration in self intoxicated patients in relation to possibly known intake of drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Sten Rubertsson, MdPhd, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
This is not applicable in this study. All patients according to protocol will be described in groups.